CLINICAL TRIAL: NCT06997315
Title: Bath MyoRhythms Project (BMP): Characterising Rhythmicity in Human Skeletal Muscle Metabolism
Brief Title: Bath Myorhythms Project
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Surrey (Other); Maastricht University (Other); University of Copenhagen (Other); University of Nottingham (Other); Australian Catholic University (Other); University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, James Betts, Professor, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 7560-9757
Record Dates: First submitted 2025-04-22; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator)
  Interventions: Other: No exercise
- Early exercise (Experimental)
  Interventions: Other: Time of exercise
- Late exercise (Experimental)
  Interventions: Other: Time of exercise

INTERVENTIONS:
Other: Time of exercise — The intervention is 1 hour of exercise at 50% between lactate threshold 1 and 2 either in the morning or the evening at the start of the 24 hour sampling period.
  Arms: Early exercise; Late exercise
Other: No exercise — The participants will rest for the full 24 hour sampling period.
  Arms: Control

SUMMARY:
Human Physiology is coordinated by a circadian timing system that synchronises daily cycles of light-dark, wake- sleep, activity-rest and feeding-fasting. The alignment of these behavioural patterns with underlying biological rhythms is closely linked to physiological function, with misalignment linked to chronic metabolic diseases.

The vast majority of evidence about rhythms in metabolism comes from studies of rodents, which is remarkable given that rodents differ fundamentally from humans in both behaviour and metabolic regulation. Moreover, almost no research in any species has examined the effects of muscle contractile activity on 24-h rhythms in metabolism. Skeletal muscle is a key site of metabolic regulation and contractile activity is a powerful stimulus to increase metabolism. The researchers have established a novel protocol for serial muscle sampling throughout 24 hours and pilot work completed in preparation for this grant revealed diurnal transcriptomic and lipidomic rhythms in human skeletal muscle. Further development of that protocol has used enteral feeding via a tube which delivers nutrient directly to the stomach to enable constant nutrient delivery (including during sleep), with preliminary data indicating that underlying rhythms in metabolism are responsive to nutrient availability patterns.

The researchers will now capitalise on those findings by incorporating multiple isotope tracers within the protocol, thus finally documenting the nature of rhythmic flux in carbohydrate metabolism and protein turnover in human skeletal muscle, and how those rhythms are aligned with timing and patterns of exercise. In summary, participants will stay in the laboratory for 36 hours with 24 hours of constant feeding via nasogastric tube, and muscle and blood sampling. Participants will be allocated to either the early or late exercise group (involving 1 hour of cycling at either 0800 or 2000 h, respectively) or the control group who will rest for the 24 hours.

DETAILED DESCRIPTION:
Once eligibility has been verified, participants will attend the laboratory for preliminary testing which will include a submaximal exercise test on an exercise bike. Participants will then be monitored for one-week ahead of their main laboratory visit and will adhere to pre-trial dietary and lifestyle controls for the final 48 h of the pre-trial week (including records of wake/sleep cycles and weighed-food diaries, along with wearable technologies to continuously monitor physical activity, light exposure and sub-cutaneous interstitial glucose concentrations) and standardised meals will be provided to all participants for the 24 h ahead of laboratory visits.

Participants will arrive in the laboratory at 1900 h (DAY 1) the day before the 24-h monitoring period to consume a standardised evening meal (baked potato, beans, broccoli). A cannula will be fitted to an antecubital vein prior and participants will sleep in the laboratory ready for monitoring to commence upon waking the next morning (DAY 2).

At 0600 h, whilst the participant remains asleep, infusion of labelled protein and glucose will be commenced to achieve steady state before starting the sampling period and to allow measurement of protein and glucose metabolism. Resting metabolic rate (the amount of energy required at rest) will be measured immediately upon waking by collecting expired breath samples. Specifically, expired gases will be collected for 20-30 minutes using the gold-standard Douglas bag technique. This measured value will then be used to individually prescribe the energy requirements to be met via nasogastric feeding. A second cannula will then be fitted and a nasogastric tube will be inserted through the nose into the stomach to commence delivery of a nutritionally balanced meal-replacement solution at 0800 h which will be delivered continuously throughout the 24 hour monitoring period. A muscle sample will be obtained at 0730. Participants in the early exercise group will commence 1 hour of exercise at a moderate intensity with 1-min expired breath samples and blood samples collected every 15 minutes and heart rate monitored throughout to verify the exercise intensity.

Further muscle samples will be obtained at 4-h intervals to allow for 7 time-points ending at the final sample at 0800 h the next morning (DAY 3) and blood sampling will occur hourly. The inactive group will follow the same sampling schedule without the exercise. The late exercise group will adhere to the same series of events as described above but with a 12-h delayed shift in time of day. Upon completion of those final tissue samples, participants will be provided with the same breakfast as they had been provided on DAY 1 as part of their dietary standardisation and they will be issued with the same lunch as was consumed on DAY 1 to take away. All wearable devices other than the continuous glucose monitor will then be removed before the participant leaves the laboratory. Body temperature will also be measured throughout the protocol via ingestible thermometers.

ELIGIBILITY:
Inclusion Criteria:

* Women and men - with targeted recruitment to encourage females to volunteer given previous recruitment rates; anticipating fewer women than men, sex will also be included as a strata in the randomisation plan to favour the few who do volunteer being relatively evenly distributed between conditions.
* A body mass index of >18 and <35 kg•m-2.
* Minimum absolute body mass of 67 kg (to accommodate the required dose of lidocaine for 7 biopsies, plus additional for pre-incisions)
* be between 18-50 years of age
* Premenopausal women
* Metabolically healthy (free from diagnosed metabolic illness or family history of type II diabetes
* be able and willing to give informed oral and written consent,
* complete and meet the defined criteria of pre-study questionnaires and screens
* have a regular sleep cycle with a sleep duration between 6 and 8 h
* do not exhibit extreme morning or evening preference (Horne and Ostberg, 1976)
* agree to keep a constant sleep/wake cycle with a self-selected 8-h duration in bed/dark trying to sleep (from which it cannot be deviated by more than 30 minutes) for one week prior to the lab study
* obtain 15 minutes of sunlight within 1.5 hours of waking up and agree to nap only within a 4 h designated nap window for one week prior to the lab study
* allow confirmation of compliance to these instructions by wearing ActiHeart and light monitors continuously and complete daily sleep and event diaries for one week before the study session
* agree to refrain from alcohol, caffeine, strenuous exercise and certain food components for one day before the study session
* agree to weigh and record daily meals (based on individual energy requirements) for TWO days prior to the study
* agree to refrain from prescribed and 'over the counter' medication and food/vitamin supplements for a wash-out period three weeks before and during the study IF the drug is deemed to affect study outcomes and may safely be withheld for that period.

Exclusion Criteria:

* are taking regular medication (also non-prescribed) or food supplements (e.g. vitamins, minerals, fish oil, antioxidant tablets) from which it is not possible to refrain, known to influence: sleep/alertness/the circadian timing system (e.g. beta-blockers, barbituates, antidepressants, benzodiazepines, melatonin, ritalin, modafinil, soporifics, St John's Wort), any of the metabolic functions (e.g. affecting thyroid, kidney, liver or gastrointestinal function) any of the inflammatory markers (e.g. aspirin, ibuprofen, antibiotics, hay fever medication, medication for sore throats and colds), and/or any of the endothelial markers (e.g. ACE inhibitors and angiotensin (receptor) blockers, diuretics, beta-blockers, anti-thrombosis medication), any anticoagulant medication
* have a history of any circadian or sleep disorder or metabolic, cardiovascular or chronic infectious / inflammatory disease as confirmed by the GP or the pre-study questionnaires (e.g. a Pittsburgh Sleep Quality Index > 5 will result in exclusion)
* have a history of psychiatric or neurological disease or drug and alcohol abuse
* have donated over 400 ml of blood in the three months preceding the study
* have participated in shift work (regularly working past a typical bed time of 2300 h) or have travelled across more than two time zones within three weeks before the study
* do not keep a regular sleep-wake cycle
* do not refrain from alcohol, caffeine containing drinks (e.g. coffee, coke, tea, Red Bull), strenuous exercise and certain foods (e.g. those high in fat and green vegetables) for one day before and during the laboratory session
* regularly consume more than 4 cups of caffeinated beverages (e.g. tea, coffee, cola) daily
* smokers
* have a known lidocaine allergy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-23 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Carbohydrate flux | 24 hours
  Rates of exogenous glucose appearance, endogenous glucose production, total carbohydrate oxidation, exogenous carbohydrate oxidation and net glycogen degradation in muscle biopsies over 24 hours
Skeletal muscle protein synthesis | 24 hours
  Plasma amino acid concentrations derived from the L-[ring-13C]-phenylalanine infusion over 24 hours.
Skeletal muscle protein synthesis | 24 hours
  Protein fractional synthetic rates in muscle samples derived from the L-[ring-13C]-phenylalanine infusion over 24 hours.
Mass spectrometry phosphoproteomics | 24 hours
  Mass spectrometry phosphoproteomics from skeletal muscle biopsies over 24 hours.
Protein content of proteins involved in insulin signalling, glucose transport and protein synthesis. | 24 hours.
  The content of proteins involved in insulin signalling, glucose transport and protein synthesis determined by semi-quantitative western blotting in skeletal muscle biopsies over 24 hours.

SECONDARY OUTCOMES:
Skeletal muscle gene expression | 24 hours
  Transcriptomic and targeted quantitative real-time PCR TaqMan analyses of skeletal muscle gene expression from muscle biopsies over 24 hours.
Intramuscular metabolites | 24 hours
  Liquid chromatography-mass spectrometry to quantify circulating and intramuscular metabolites indicative of carbohydrate, lipid and amino acid metabolism in skeletal muscle biopsies over 24 hours.
Intramuscular enzymes | 24 hours
  Liquid chromatography-mass spectrometry to quantify the activation of intramuscular enzymes involved in the formation of acetyl-CoA in skeletal muscle biopsies over 24 hours.
Plasma glucose concentrations | 24 hours
  Plasma glucose concentrations over 24 hours.
Plasma non-esterified fatty acid concentrations | 24 hours
  Plasma non-esterified fatty acid concentrations over 24 hours
Plasma glycerol concentrations | 24 hours
  Plasma glycerol concentrations over 24 hours
Plasma triacylglycerol concentrations | 24 hours
  Plasma triacylglycerol concentrations over 24 hours
Plasma urea concentrations | 24 hours
  Plasma urea concentrations over 24 hours
Plasma insulin concentrations | 24 hours
  Plasma insulin concentrations over 24 hours
Plasma glucagon-like peptide-1 concentrations | 24 hours
  Plasma glucagon-like peptide-1 concentrations over 24 hours
Plasma insulin-like growth factor 1 concentrations | 24 hours
  Plasma insulin-like growth factor 1 concentrations over 24 hours
Plasma gastric inhibitory polypeptide concentrations | 24 hours
  Plasma gastric inhibitory polypeptide concentrations over 24 hours
Plasma peptide YY concentrations | 24 hours
  Plasma peptide YY concentrations over 24 hours
Plasma cortisol concentrations | 24 hours
  Plasma cortisol concentrations over 24 hours
Plasma total ghrelin concentrations | 24 hours
  Plasma total ghrelin concentrations over 24 hours
Plasma leptin concentrations | 24 hours
  Plasma leptin concentrations over 24 hours
Plasma melatonin concentrations | 24 hours
  Plasma melatonin concentrations over 24 hours

OTHER OUTCOMES:
Skeletal muscle lipid concentrations | 24 hours
  Skeletal muscle lipid concentrations using lipidomics of muscle biopsy samples over 24 hours
Blood cell counts | 24 hours
  Plasma blood cell counts (i.e. leukocytes and subsets, erythrocytes and platelets) over 24 hours.
Skeletal muscle autophagic flux | 24 hours
  Protein content of proteins involved in skeletal muscle autophagic flux determined by semi-quantitative western blotting in muscle biopsy samples over 24 hours.
Polysomnography profile | 11 hours
  During 11 hours of sleep during pre-trial monitoring and intervention.
Heart rate during exercise | 60 minutes
  Bpm
Rate of perceived exertion during exercise | 60 minutes
  Borg scale
Body temperature | 24 hours
  Body temperature over 24 hours
Blood pressure | 24 hours
  Blood pressure over 24 hours, mmHg.
Energy expenditure during exercise | 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes